CLINICAL TRIAL: NCT03526432
Title: A Phase II, Single Arm Study of Atezolizumab + Bevacizumab in Women With Advanced, Recurrent or Persistent Endometrial Cancer
Brief Title: Phase II Study of Atezolizumab + Bevacizumab in Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-GEN-001
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bevacizumab + Atezolizumab (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at 15mg/kg on Day 1 of every 21-days cycle.
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until disease progression, unacceptable toxicity, loss of clinical benefit as determined by the investigator.

SUMMARY:
This is a single arm, Phase II study using the combination of atezolizumab and bevicacizumab in women with advanced, recurrent or persistent endometrial cancer. Safety and futility of this drug combination will be assessed to see what effect this treatment has on this patient population.

DETAILED DESCRIPTION:
This phase 2 study using atezolizumab and bevacizumab aims to study the objective tumor response in women with recurrent endometrial cancer. Drugs will be administered via IV every 21 days until disease progression, unacceptable toxicity, or loss of clinical benefit as determined by investigator. Subjects will receive routine cancer care as well as tests and procedures required for the purposes of this study. It is expected this combination will be produce an anti-cancer effect with manageable toxicities in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of endometrial carcinoma (including endometrioid, serous, mixed adenocarcinoma, clear-cell carcinoma, or carcinosarcoma).
2. Evidence that the endometrial cancer is advanced, recurrent, or persistent and has relapsed or is refractory to curative therapy or established treatments.
3. At least 1 prior platinum-based chemotherapeutic regimen, but not more than 2 prior chemotherapeutic regimens, for management of endometrial carcinoma. Prior treatment may include chemotherapy, and/or consolidation/maintenance therapy.
4. Measurable disease by RECIST 1.1, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm in long axis when measured by CT, MRI, or caliper measurement by clinical exam. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI.
5. Female patients 18 years or older.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
7. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods as defined in study protocol.
8. Clinical laboratory values as specified in study protocol within 4 weeks before the first dose of study drug.
9. Able to understand and willing to sign the Informed Consent Form and the written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
10. Must have ability to comply with the study protocol, in the investigator's judgment.
11. Patients MSI status must be known (via immunohistochemistry)
12. Patients should have archival tumor tissue available or agree to have pre-treatment tumor biopsy if no archival tissue is available for correlative studies If unable to be safely biopsied and patient desires enrollment, may be enrolled per principal investigator discretion.
13. Life expectancy of greater than 12 weeks.

Exclusion Criteria:

1. Positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug. Women who are lactating and breast feeding are not eligible.
2. Previous treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody.
3. History of auto-immune disorders (SLE, sarcoidosis, RA, Crohn's).
4. Initiation of treatment with systemic corticosteroids (either IV or oral steroids, excluding inhalers) within 1 week before administration of the first dose of study drug
5. Sensory or motor neuropathy ≥ Grade 2.
6. Patients with symptomatic, untreated Central nervous system (CNS) metastasis; Patients with a history of treated CNS lesions are eligible if all criteria provided per study protocol are met.
7. Other clinically significant co-morbidities, such as uncontrolled pulmonary disease, active CNS disease, severe cardiac disease, bleeding diathesis, active infection, or any other condition that could compromise participation of the patient in the study.
8. Diagnosed or treated for another malignancy within 2 years before administration of the first dose of study drug or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
9. Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
10. Patients who have had investigational therapy, chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (other than alopecia) due to agents administered more than 4 weeks earlier; however, some therapies are allowed per study protocol.
11. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to cycle 1, day 1
12. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, compounds similar to bevacizumab or atezolizumab, or Chinese hamster ovary products.
13. Major surgical procedure within 28 days prior to cycle 1, day 1 or anticipation of need for a major surgical procedure during the course of the study
14. History of abdominal/pelvic fistula, gastrointestinal perforation and/or intraabdominal abscess within 6 months prior to day 1. Serious or non-healing wound, active ulcer or bone fracture
15. Immunocompromised patients and subjects known to be HIV positive and currently receiving antiretroviral therapy. NOTE: Subjects known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience complete or partial tumor response | 3 years
  To estimate the objective tumor response in women of this patient population

SECONDARY OUTCOMES:
Progression-free Survival | up to 3 years
  To estimate progression-free survival (PFS) and overall survival (OS) of patients with recurrent or persistent endometrial cancer treated with Atezolizumab and Bevacizumab.
Overall survival | up to 3 years
  To estimate overall survival (OS) of patients with recurrent or persistent endometrial cancer treated with Atezolizumab and Bevacizumab.
Number of patients who experience toxicity | 6 months
  To determine the nature and degree of toxicity in combination of atezolizumab and bevacizumab.
Number of participants who experience immune related response | 6 months
  To estimate response using immune related response criteria (irRC) in patients receiving Atezolizumab and Bevacizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, MD, Principal Investigator — Obstetrics and Gynecology
Locations (3):
- United States (3):
  - UAB Women and Infants Center, Birmingham, Alabama
  - Washington University School of Medicine, St Louis, Missouri
  - Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No